CLINICAL TRIAL: NCT06508801
Title: Blood Flow Restriction for Optimizing Balance in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Anjali Sivaramakrishnan, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00000472BFR; P30AG044271 (NIH)
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: Blood flow restriction; Instability resistance training; Balance; Strength; Postural control
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Two group, randomized, repeated measure design
Who Masked: Participant, Investigator
Masking Description: This study will utilize block randomization with permuted blocks in a 1:1 ratio. Individuals will be assigned to either Group 1 or Group 2 after baseline assessment. The randomization will be predetermined, and the allocation will be concealed. Only the statistician and research coordinator will be aware of the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFR plus IRT Group (Experimental): Blood Flow Restriction plus Instability Resistance Training group. Participants will receive 2 sessions per week over 6 weeks.
  Interventions: Other: Blood flow restriction training; Other: Instability Resistance Training
- IRT Only Control Group (Other): Instability Resistance Training only group. Participants will receive 2 sessions per week over 6 weeks.
  Interventions: Other: Instability Resistance Training

INTERVENTIONS:
Other: Blood flow restriction training — The BFR Intervention will consist of 75 repetitions; reps (set 1: 30 reps, sets 2 - 4: 15 reps with 30 s of rest between sets and 1 minute between exercises) at 20-30% of 10 repetition maximum (RM). BFR training will be performed during toe raises, lunges and single leg stance exercises on unstable surfaces (i.e., foam, Dyna disc, balance disc, and BOSU-ball®) as tolerated by the participant.
  Other Names: BFR
  Arms: BFR plus IRT Group
Other: Instability Resistance Training — The following devices will be used for instability training: foam, dyna disc, balance disc and BOSU-ball®. Unstable devices will be changed during the six-week period from the least to the most unstable devices. Once a participant reduces the body sway on a device, the device will be progressed. Participants will perform IRT with or without blood flow restriction.
  Other Names: IRT

SUMMARY:
This study is being done to understand how reducing blood flow (BRT) during balance-challenging strengthening exercises (instability resistance training, or IRT) can help improve symptoms of Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a disease of the nervous system that attacks the nerve cells in the brain responsible for controlling movement in the arms, legs and face. It is a progressive condition that gets worse with time. The purpose of this study is to determine the effects of blood flow restriction (BFR) in combination with strengthening exercises that challenge balance (instability resistance training (IRT)) to improve the symptoms of the participant's condition. This research is being done to understand the effects of BFR with IRT on symptoms of PD such as balance, mobility, walking and endurance. There will be two groups 1 and 2; group 1 will perform IRT with BFR and group 2 will perform IRT only. Each session with either intervention will last approximately 45 minutes. Researchers will test the effects of the intervention on the participant's walking ability, balance function and endurance. The researchers hope to learn whether low resistance exercises using these tight cuffs around the thighs are well tolerated by individuals with PD and determine whether there is an improvement in muscle strength, balance, and physical function. In addition, researchers will also use peripheral nerve stimulation techniques which are non-invasive (does not go inside the body). These techniques will be used to measure spinal excitability (i.e., nerve stimulator for testing strength of the pathway between spinal cord and muscles) in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages 40 - 85 with a diagnosis of idiopathic Parkinson's Disease (PD) consistent with the United Kingdom PD society brain bank criteria,
2. in Hoehn and Yahr stage 2-4,
3. a score of ≥23 on the mini-Mental Scale Examination.

Exclusion Criteria:

1. History of cardiovascular disease, uncontrolled hypertension (blood pressure ≥140/90 mmHg), orthostatic hypotension, deep-vein thrombosis, varicose veins, or rhabdomyolysis;
2. Ankle branchial index ≤ 0.9 or > 1.3.
3. History of other neurological disorders affecting the central nervous system such as stroke, multiple sclerosis, tumors, amyotrophic lateral sclerosis or muscle disease such as muscular dystrophy, myopathy.
4. History of uncontrolled diabetes, severe osteoporosis, or cognitive impairment.
5. Body mass index above 40; such individuals are more likely to have poorer muscle function and more pain.
6. Absolute contraindications to exercise as per the American College of Sports Medicine (uncontrolled arrhythmias, third-degree heart block, recent electrocardiogram (EKG) changes, unstable angina, acute myocardial infarction, or acute congestive heart failure
7. Had surgery in the lower extremities within the past 6 months.
8. Pre-menopausal and not on birth control
9. Pregnant or planning to become pregnant within the course of the study
10. Plan to have major surgery within 2 months.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility metric | Baseline to 6 weeks
  The treatment will be considered acceptable if the dropout and significant adverse event rate is less than 20%, that is no more than 2 out of 10 participants in the treatment group either 1) drop out, 2) withdraw consent, or 3) have a significant adverse event (Grade 3 or higher on 5 point scale where 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = death). Results will be reported as percentage of participants that dropped out.

SECONDARY OUTCOMES:
Balance Measure | Baseline to 14 weeks
  Balance will be measured using the miniBESTest Balance Evaluation Systems Test. The test has a range of scores from 0 to 28 points from 14 items that are each scored from 0-2.
  "0" indicates the lowest level of function and "2" the highest level of function. Equipment used: Temper® foam (also called T-foamTM 4 inches thick, medium density T41 firmness rating), chair without arm rests or wheels, incline ramp, stopwatch, a box (9" height) and a 3 meter distance measured out and marked on the floor with tape [from chair].
Functional Mobility | Baseline to14 weeks
  The 30-second chair stand (30CST) will be used to assess functional mobility. In this test a person needs to stand up from sitting as many times as possible in 30 seconds. An increase in the number of stands is suggestive of better lower extremity strength
Movement Disorder Society Unified Parkinson's Disease Rating Scale | Baseline to 14 weeks
  Motor severity will be assessed by the Movement Disorders Society - Unified Parkinson's Disease Rating Scale - part III. This scale is the gold standard for measuring the severity and progression of PD. Part III entails motor examination which consists of 18 questions that are scored on a 0-4 scale with a total score range between 0 and 72. Higher scores suggest greater severity and progressing disease.
Postural Sway (Biosway) | Baseline to 14 weeks
  Participants will perform postural sway assessments on the Biodex BioSway. Participants will maintain a consistent foot position which will be recorded and kept constant for all trials. Change in postural stability will be compared from baseline to follow up assessments.
Spinal Excitability Assessment | Baseline to 14 weeks
  Spinal reflex excitability will be measured by eliciting the H-reflex. Subjects will lay down in a prone position. Surface recording electrodes will be placed over the soleus muscle. The tibial nerve will be stimulated with a nerve stimulator. The reference electrode would be placed over the knee cap. Once stimulation electrodes are positioned, H-reflex and M-wave recruitment curves will be obtained. Stimulus intensity will be increased every 5 seconds by 2 mA increments until the maximum H-reflex (Hmax) is obtained and then increased by 10 mA increments until the maximal M response is obtained (Mmax). The M-wave target amplitude will be monitored to ensure stability of stimulation throughout the experiment while eliciting an H-reflex recruitment curve. The H wave amplitude will be expressed as a % of the Mmax (maximum M wave) amplitude.
Hip abductor muscle strength | Baseline to 14 weeks
  Muscle strength for hip abductors will be measured with isokinetic dynamometry.
Knee extensor muscle strength | Baseline to 14 weeks
  Muscle strength for knee extensors will be measured with isokinetic dynamometry.
Ankle plantar flexor muscle strength | Baseline to 14 weeks
  Muscle strength for ankle plantar flexors will be measured with isokinetic dynamometry.
Quality of Life PDQ-39 Questionnaire | Baseline to 14 weeks
  The Parkinson's Disease Questionnaire (PDQ)-39 is a widely used tool for evaluating quality of life in PD. It consists of 39 items that cover seven domains such as mobility, activities of daily living, emotional well-being, stigma, social support, cognition, and communication. Scores on each item range from 0-4 with 0 indicating never and 4 indicating always. These scores are converted to a summary index score which ranges from 0 - 100, with lower scores suggesting higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Sivaramakrishnan, PhD, PT, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected Individual Participant Data (IPD), all IPD that underlie results in a publication will be shared with colleagues.
Supporting Information: SAP, ICF
Time Frame: At the time of publication in a peer review journal